CLINICAL TRIAL: NCT00175981
Title: Pharmacokinetic and Pharmacodynamic Evaluation of the Interaction Between Fluvoxamine and Sildenafil in Healthy Males
Brief Title: Interaction Between Fluvoxamine and Sildenafil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: K058
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Healthy
MeSH Terms: interventions — Sildenafil Citrate; Fluvoxamine

INTERVENTIONS:
Drug: sildenafil, fluvoxamine

SUMMARY:
Aim of the study is to assess the interaction between sildenafil and fluvoxamine and its effect on the venous response to sodium nitroprusside.

DETAILED DESCRIPTION:
In a randomised, double-blind, placebo-controlled, cross-over study in healthy men we will assess the effect of oral fluvoxamine (50mg qd on day 1-3; 100mg qd on day 4-10) on sildenafil kinetics (single oral 50mg dose on day 11). Sildenafil plasma concentrations will be determined by LC/MS. We will also assess the effect of sildenafil on venodilation induced by a constant dose-rate of the NO-donor sodium nitroprusside (SNP) during preconstriction with phenylephrine (dorsal hand vein compliance technique).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male individuals, age: 18-45.
* Able and willing to give written informed consent

Exclusion Criteria:

* Hypotension ( 65 mmHg diastolic and  100 mmHg systolic blood pressure)
* Bleeding disorders in medical history
* Intake of medication impairing platelet function or influencing coagulation (for example aspirin, NSAID and others) during the preceding 4 weeks
* Known condition causing endothelial dysfunction (e.g. diabetes, hyperlipidaemia, arterial hypertension, hyperhomocysteinaemia, smoking)
* Anatomic deformity of the penis like angulation, penile fibromatosis (peyronie's disease) or diseases favouring priapism (e.g. leukaemia, plasmocytoma, sickle-cell anaemia)
* Regular medication and/or treatment with drugs within the preceding 4-6 weeks (exclusion has to be decided in each case)
* alcohol (>30 g/d) or drug abuse
* Acute or chronic illness
* Blood donation within the preceding 2 months
* Participation in clinical trial within 2 month before the study
* Drug and/or alcohol abuse.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2003-02; Study Completion 2004-11

PRIMARY OUTCOMES:
Drug-induced changes of hand vein compliance
Drug-induced changes of pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Walter E Haefeli, MD, Principal Investigator — Heidelberg University
Locations (1):
- Dept. of Internal Medicine VI, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany